CLINICAL TRIAL: NCT01288950
Title: Vitamin D Supplementation Enhances Immune Response to BCG Vaccination in Infants
Brief Title: Vitamin D Supplementation Enhances Immune Response to Bacille-Calmette-Guerin (BCG) Vaccination in Infants
Acronym: BCG-25-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Principal Investigator, Amaran Moodley, Research Fellow, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NR-0138
Record Dates: First submitted 2011-02-01; First posted 2011-02-03 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-08

CONDITIONS: Tuberculosis
Keywords: BCG vaccine; Vitamin D; Cholecalciferol; Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D3 (Experimental)
  Interventions: Dietary Supplement: Vitamin D3 (cholecalciferol)
- Placebo (No Intervention)

INTERVENTIONS:
Dietary Supplement: Vitamin D3 (cholecalciferol) — A single oral dose of 50,000 IU of vitamin D3 (cholecalciferol) will be given prior to Bacille-Calmette-Guerin (BCG) vaccination
  Other Names: Carlson Ddrops liquid vitamin D3 2,000 IU per drop
  Arms: Vitamin D3

SUMMARY:
The purpose of this study is to determine whether a single oral dose of vitamin D given to infants prior to Bacille-Calmette-Guerin (BCG) vaccination will enhance the immune response to BCG vaccination.

DETAILED DESCRIPTION:
In 2000, there were an estimated 884,000 cases of tuberculosis (TB) in children with many developing severe, disseminated disease. Widespread immunization with Bacille-Calmette-Guerin (BCG) vaccine has not been effective in preventing primary TB infection or in halting the progression from latent to active disease. Poor vaccine efficacy has prompted investigators to develop novel TB vaccines and to experiment with enhancing the immune response to the current BCG vaccine.

Increasing data indicate that children with low vitamin D levels and specific genetic variants that lower functional levels of vitamin D are at increased risk for severe tuberculosis. Elegant studies investigating Mycobacterium tuberculosis (Mtb) infection have shown that mycobacteria are able to reside in endosomes within macrophages by preventing endosome-lysosome fusion; a critical step in autophagy, a cellular process used to recycle cytoplasmic organelles and proteins, and to degrade microbial organisms including Mtb. In-vitro studies have shown that vitamin D increases autophagy and triggers the production of antimicrobial peptides including cathelicidin. This leads to increased intracellular killing of Mtb and increased Mtb antigen presentation to the immune system. Anti-tuberculous vaccines that over-express Mtb antigens generate a stronger immune response than wild type BCG vaccine.

The investigators hypothesis is that a single oral dose of vitamin D3 (cholecalciferol) given to infants prior to BCG administration will enhance the immune response to vaccination through improved MHC class I and class II presentation of the vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy mothers > 18 years of age
* Term, healthy infants eligible to receive the Bacille-Calmette- Guerin (BCG) vaccine

Exclusion Criteria:

* Recent maternal history of tuberculosis (within 1 year) or active tuberculosis
* Known maternal human immuno-deficiency virus (HIV) infection
* Maternal fever or chorio-amnionitis
* Maternal use of vitamin D, steroids or immuno-regulatory medications
* Household member with active tuberculosis

Max Age: 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2011-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Bacille-Calmette-Guerin (BCG) vaccine efficacy | 2 months
  BCG vaccine efficacy will be assessed by measuring the host immune response against BCG at 2 months, 6 months and one year after BCG immunization. A whole blood assay will be used to measure multiple cytokines and mycobacterial growth suppression.
Bacille-Calmette-Guerin (BCG) vaccine efficacy | 6 months
Bacille-Calmette-Guerin (BCG) vaccine efficacy | 1 year

SECONDARY OUTCOMES:
Effect of a single dose of 50,000 IU vitamin D3 on serum vitamin D levels | 2 months
  Serum 25 hydroxy (OH) vitamin D levels will be measured prior to vitamin D supplementation and at 2 months, 6 months and one year after BCG immunization. The investigators will also determine whether specific host genetic variants including the Fok-I(rs2228570T/C), Bsm-I(rs1544410A/G), GC(rs2282679A/C), DHCR7(rs12785878G/T) and CYP2R1 (rs10741657A/G) polymorphisms affect baseline vitamin D levels and alter the response to vitamin D supplementation.
Bacille-Calmette-Guerin (BCG) vaccine efficacy | 1 year
  The investigators will determine whether specific host genetic variants including the Fok-I(rs2228570T/C), Bsm-I(rs1544410A/G), GC(rs2282679A/C), DHCR7(rs12785878G/T) and CYP2R1 (rs10741657A/G) polymorphisms affect the response to BCG vaccine in infants receiving either vitamin D or placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Spector, MD, Study Chair — University of California, San Diego; Amaran Moodley, M.D, Principal Investigator — University of California, San Diego
Locations (1):
- Tijuana General Hospital, Tijuana, Estado de Baja California, Mexico

REFERENCES:
- [Derived] Huey SL, Acharya N, Silver A, Sheni R, Yu EA, Pena-Rosas JP, Mehta S. Effects of oral vitamin D supplementation on linear growth and other health outcomes among children under five years of age. Cochrane Database Syst Rev. 2020 Dec 8;12(12):CD012875. doi: 10.1002/14651858.CD012875.pub2. PMID 33305842